CLINICAL TRIAL: NCT01242605
Title: ABC-04 a Phase 1B Study of Cisplatin, Gemcitabine and Selumetinib in Patients With Advanced Biliary Tract Cancer
Brief Title: ABC-04 a Study of Cisplatin, Gemcitabine and Selumetinib in Patients With Advanced Biliary Tract Cancer
Acronym: ABC-04
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/10/0254; 2010-018522-39 (EudraCT Number)
Record Dates: First submitted 2010-07-06; First posted 2010-11-17 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2015-10

CONDITIONS: Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms
Keywords: unresectable; advanced
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — AZD 6244; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single armed (Experimental): This is not a randomised trial, there is only one study group. All patients will receive cisplatin/gemcitabine chemotherapy in addition to oral daily dosing of selumetinib
  Interventions: Drug: selumetinib; Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: selumetinib — The starting dose of selumetinib will depend on the cohort. The first dose of selumetinib to be studied will be 75 mg twice daily (bd). Selumetinib will be taken every day (continuously) either once or twice a day, depending on the dose. Treatment with selumetinib may continue until disease progression.
  Other Names: AZD6244
Drug: gemcitabine — gemcitabine: taken in combination with cisplatin will be given at 1000 mg/m*2 in 250 - 500 ml 0.9% saline over 30 minutes by intravenous infusion on days 1, and 8 of each 21-day cycle for eight cycles in total
Drug: cisplatin — cisplatin: 25 mg/m*2 in 1000 ml 0.9% saline given over 1 hour followed by 500mls 0.9% saline over 30 minutes followed by gemcitabine on days 1, and 8 of each 21-day cycle for eight cycles in total

SUMMARY:
The objective of this study is to establish the recommended dose of selumetinib, a novel MEK inhibitor for use in combination with gemcitabine and cisplatin.

DETAILED DESCRIPTION:
This trial aims to evaluate the safety and tolerability of selumetinib in combination with CisGem and to establish the recommended dose to take into phase II studies. Pharmacokinetic and pharmacodynamic endpoints will be assessed and preliminary efficacy data will also be collected.

Patients with Advanced Biliary tract Cancer will receive CisGem regimen and selumetinib. A dose de-escalation scheme will be employed to determine the recommended phase II dose of selumetinib.

Patients will be recruited in cohorts of three and assessed for dose limiting toxicity (DLT) during the first cycle of treatment. Depending on the number of DLTs observed, the cohort may be expanded, the next cohort may be enrolled at a lower dose or the dose may be declared the recommended dose. Patients will receive up to eight cycles of CisGem and may continue to receive selumetinib until progression of disease.

ELIGIBILITY:
Inclusion Criteria:

* A histopathological or cytological diagnosis of non-resectable, recurrent or metastatic biliary tract (intra- or extra-hepatic), gallbladder or ampullary carcinoma
* ECOG performance status 0, 1, or 2
* Age ≥ 18
* Estimated life expectancy > 3 months
* Adequate haematological function:

  * Haemoglobin 9g/dL (prior transfusions for patients with low haemoglobin are allowed)
  * WBC >/= 3.0 x 10*9/L
  * Absolute neutrophil count (ANC) >/= 1.5 x 10*9/L
  * Platelet count >/= 100 x 10*9/L
* Adequate liver function:

  * Total bilirubin ≤1.5 x upper limit of normal (ULN) OR ≤ 3.0 x upper limit of normal (ULN) if stable for a duration of two weeks
  * ALT and/or AST & alkaline phosphatase ≤ 5 x ULN
* Adequate renal function:

  * Serum urea and serum creatinine < 1.5 times ULN
  * Calculated GFR >/= 45 mL/min. If the calculated GFR is below 45ml/min, isotope EDTA confirmation of adequate renal function is required
* Capable of giving written informed consent
* Prior therapy is allowed (provided there has been a full recovery):

  * Surgery (non-curative operation), must have evidence on nonresectable disaes progression prior to trial entry
  * Radiotherapy, must have clear evidence of disease progression prior to inclusion
  * Prior adjuvant chemotherapy is allowed provided neither gemcitabine nor cisplation were used and treatment was completed 28 days prior to trial entry.

Exclusion Criteria:

* Any prior exposure to MEK, Ras, or Raf inhibitors
* Cardiac conditions as follows:

  * Uncontrolled hypertension (BP ≥150/95 despite optimal therapy)
  * Heart failure (NYHA Class II or above)
  * Prior or current cardiomyopathy
  * Baseline LVEF ≤50%
  * Atrial fibrillation with heart rate >100 bpm
  * Unstable ischaemic heart disease (MI within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly).
* Incomplete recovery from previous surgery.
* Patients undergoing current treatment with curative intent.
* History of prior malignancy that could interfere with the response evaluation (exceptions include in-situ carcinoma of the cervix treated by cone-biopsy/resection, non-metastatic basal and/or squamous cell carcinomas of the skin, any early stage (stage I) malignancy adequately resected for cure greater than 5 years previously).
* Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial.
* Any psychiatric or other disorder (e.g brain metastases) likely to impact on informed consent.
* Pregnancy or breast-feeding. Women of child-bearing potential should must have a negative pregnancy test prior to study entry AND be using an adequate contraception method, which must be continued for 3 months after completion of chemotherapy
* NB. Whilst not excluded, patients with significant impaired hearing must be made aware of potential ototoxicity and may choose not to be included. If included, baseline audiograms are recommended and should be followed by repeat audiograms prior to cycle 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of the combination of cisplatin, gemcitabine and selumetinib, and to establish the recommended phase II dose of selumetinib when given in this combination. | from baseline to 28 days post last patient last treatment
  To investigate the safety and tolerability of the combination of cisplatin, gemcitabine (CisGem) and selumetinib and to establish the recommended phase II dose of selumetinib when given in this combination.
  The recommended dose of selumetinib to use in combination with CisGem in future studies will be the dose at which less than 33% of patients experience a DLT. The recommended dose will not be higher than 75mg/m*2

SECONDARY OUTCOMES:
Response rate | From baseline to end of treatment
  To make a preliminary assessment of efficacy in terms of tumour control.

CONTACTS AND LOCATIONS:
Overall Officials: John Bridgewater, MBBS, Principal Investigator — UCL
Locations (3):
- United Kingdom (3):
  - Hammersmith Hospital, London
  - University College London Hospital, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bridgewater J, Lopes A, Beare S, Duggan M, Lee D, Ricamara M, McEntee D, Sukumaran A, Wasan H, Valle JW. A phase 1b study of Selumetinib in combination with Cisplatin and Gemcitabine in advanced or metastatic biliary tract cancer: the ABC-04 study. BMC Cancer. 2016 Feb 24;16:153. doi: 10.1186/s12885-016-2174-8. PMID 26912134
- See also: Publication — http://bmccancer.biomedcentral.com/articles/10.1186/s12885-016-2174-8